CLINICAL TRIAL: NCT04646109
Title: The Effectiveness and Safety of Ivermectin as add-on Therapy in Severe COVID-19 Management
Brief Title: Ivermectin for Severe COVID-19 Management
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Collaborators: NeuTec Pharma (Industry)
Responsible Party: Principal Investigator, Nurullah Okumuş, Prof. Dr., Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IVMC_03
Record Dates: First submitted 2020-11-15; First posted 2020-11-27 (Actual); Results first posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: COVID-19
Keywords: Ivermectin; SARS-CoV-2; Treatment
MeSH Terms: conditions — COVID-19 | interventions — Ivermectin; Hydroxychloroquine; favipiravir; Azithromycin

STUDY DESIGN:
Intervention Model Description: Patients who were hospitalised with a pre-diagnosis of severe COVID-19 pneumonia and thereafter diagnosis of COVID-19 was also confirmed microbiologically with polymerase chain reaction (PCR) positivity in respiratory tract samples were included into the study. They were randomized to the study and control group, respectively. Single numbered patients were accepted as study group and double numbered patients as control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): Patients who were hospitalised with a pre-diagnosis of severe COVID-19 pneumonia and thereafter diagnosis of COVID-19 was also confirmed microbiologically with PCR positivity in respiratory tract samples were included into the study. They were randomized to the control and study group, respectively. Hydroxychloroquine, favipiravir and azithromycin (HFA) standard treatment protocol were given to the control group as recommended in the "COVID-19 (SARS-CoV-2 Infection) Guide" prepared by the Republic of Turkey Ministry of Health.
- Study Group (Experimental): In addition to HFA treatment, ivermectin 200 micrograms/kg/day (9mg between 36-50 kg, 12mg between 51-65 kg, 15mg between 66-79 kg and 200 micrograms/kg in > 80 kg) in the form of a solution prepared for enteral use was added (HFA+I) to the treatment protocol of the study group's for five days. Blood sample was taken with the first dose of ivermectin and haplotype analysis was performed in ABCB1 and CYP3A4 genes in the whole study group.
  Interventions: Drug: Ivermectin

INTERVENTIONS:
Drug: Ivermectin — Ivermectin 5mg/5ml solution was manufactured by NEUTEC™ Pharmaceutical Company-Turkey, under "Good Manufacturing Practices" (GMP) certification conditions.
  Other Names: Hydroxychloroquine, favipiravir and azithromycin
  Arms: Study Group

SUMMARY:
In this multicenter study; it was aimed to investigate the effectiveness and safety of ivermectin use in the treatment of patients with severe COVID-19 pneumonia that have no mutations which alter ivermectin metabolism and cause side effects.

DETAILED DESCRIPTION:
Patients with severe COVID-19 pneumonia were included in the study. Two groups, the study group and the control group, took part in the study.

Ivermectin 200 mcg/kg/day for five days (9 mg between 36-50 kg, 12 mg between 51-65 kg, 15 mg between 66-79 kg and 200 microgram/kg in > 80 kg) in the form of a solution prepared for enteral use added to the reference treatment protocol -hydroxychloroquine (2x400mg loading dose followed by 2x200mg, po, 5 days) + favipiravir (2x1600mg loading dose followed by 2x600mg maintenance dose, po, total 5 days) + azithromycin (first day 500mg followed by 4 days 250mg/day, po, total 5 days)- of patients included in the study group. Patients in the control group were given only reference treatment with 3 other drugs without ivermectin.

The mutations in 29 pairs of primers in mdr1/abcab1 gene by sequencing analysis using Sanger method, and the haplotypes and mutations of the CYP3A4 gene that cause the function losing were investigated among the patients who meet criteria and who were included in the study group according to randomization. Mutation screening was done when the first dose of the research drug ivermectin was given, ivermectin treatment was not continued in patients with mutations detected as a result of genetic examination and these patients were excluded from the study.

Patients were followed for 5 additional days after treatment. At the end of the treatment and follow-up period (At the end of 10th day), clinical response and changes in oxygenation and laboratory parameters were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were hospitalised with a pre-diagnosis of "severe COVID-19 pneumonia" and thereafter diagnosis of COVID-19 was also confirmed microbiologically with PCR positivity in respiratory tract samples were included into the study. They were randomized to the study and control group, respectively.

Patients with at least one of the criteria below were accepted as patients with severe COVID-19 pneumonia;

1. Presence of tachypnea ≥ 30/minute, SpO2 level < 90% in room air, PaO2/FiO2 <300 in oxygen receiving patient
2. Presence of specific radiological finding for COVID-19 in lung tomography (bilateral lobular, peripherally located, diffuse patchy ground glass opacities)
3. Mechanical ventilation requirement
4. Acute organ dysfunction findings; patients with SOFA (sepsis-related organ failure assessment) score >2

Exclusion Criteria:

* Patients with the following characteristics were excluded from the study.

  1. Pediatric patients; <18 years of old
  2. Patients with chronic liver or kidney disease
  3. Pregnant women
  4. Patients with known ivermectin allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2020-09-02 (Actual); Study Completion 2020-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nurullah Okumuş, Prof. Dr., Study Chair — Afyonkarahisar Health Science University, Afyonkarahisar, Turkey; Neşe Demirtürk, A. Prof. Dr., Study Director — Afyonkarahisar Health Science University, Afyonkarahisar, Turkey; Rıza A. Çetinkaya, Prof. Dr., Study Director — Haydarpasa Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey; Rahmet Güner, Prof. Dr., Study Director — Yıldırım Beyazıt University, Ankara City Hospital, Ankara, Turkey; İsmail Y. Avcı, Study Director — Gulhane Faculty of Medicine, University of Health Sciences, Ankara, Turkey
Locations (4):
- Turkey (Türkiye) (4):
  - Afyonkarahisar Health Science University, Afyonkarahisar
  - Gulhane Faculty of Medicine, University of Health Sciences, Ankara
  - Yıldırım Beyazıt University, Ankara City Hospital, Ankara
  - Haydarpasa Sultan Abdulhamid Han Training and Research Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Jean SS, Lee PI, Hsueh PR. Treatment options for COVID-19: The reality and challenges. J Microbiol Immunol Infect. 2020 Jun;53(3):436-443. doi: 10.1016/j.jmii.2020.03.034. Epub 2020 Apr 4. PMID 32307245
- [Background] Croci R, Bottaro E, Chan KW, Watanabe S, Pezzullo M, Mastrangelo E, Nastruzzi C. Liposomal Systems as Nanocarriers for the Antiviral Agent Ivermectin. Int J Biomater. 2016;2016:8043983. doi: 10.1155/2016/8043983. Epub 2016 May 8. PMID 27242902
- [Background] Heidary F, Gharebaghi R. Ivermectin: a systematic review from antiviral effects to COVID-19 complementary regimen. J Antibiot (Tokyo). 2020 Sep;73(9):593-602. doi: 10.1038/s41429-020-0336-z. Epub 2020 Jun 12. PMID 32533071
- [Background] Caly L, Druce JD, Catton MG, Jans DA, Wagstaff KM. The FDA-approved drug ivermectin inhibits the replication of SARS-CoV-2 in vitro. Antiviral Res. 2020 Jun;178:104787. doi: 10.1016/j.antiviral.2020.104787. Epub 2020 Apr 3. PMID 32251768
- See also: World Health Organization (WHO) Coronavirus Disease (COVID-19) Dashboard — https://covid19.who.int/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: At the beginning of the study, it was planned to have 30 patients each in the control and study groups. During the study, 6 patients were excluded from the study group because ivermectin treatments were terminated due to the detection of mutations that impairs ivermectin metabolism and new patients were added. As a result, 66 patients were included in the study, 6 patients were excluded due to mutation detection and the study was completed with 30 patients in both groups.
Period: Overall Study
Arm/Group | Control Group | Study Group
Started | 30 | 36
Completed | 30 | 30
Not Completed | 0 | 6
Not completed — Mutation disrupting ivermectin metabolism was found in 6 patients | 0 | 6

BASELINE CHARACTERISTICS:
Population: 36 patients were included in the study group. But, 6 patients in the study group were excluded from the study and analysis because ivermectin treatments were terminated due to the detection of a mutation that impairs ivermectin metabolism. As a result, overall number of baseline participants in the study group was 30.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Study Group | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Customized [Mean (Standard Deviation); unit: years] | 66.23 (13.31) | 58.17 (11.52) | 62.20 (13.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 19 | 21 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 30 | 30 | 60
Region of Enrollment [Number; unit: participants]
  Turkey | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Gender Distribution of the Patients
Description: The gender of patients (Male/female) in both groups were recorded at the time of inclusion.
Time Frame: At the first day of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 30 | 30
Participants
  Male | 19 | 21
  Female | 11 | 9

2. Primary Outcome: Age Distribution of the Patients
Description: The age of the patients (years) in both groups were recorded at the time of inclusion.
Time Frame: At the first day of the study
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 30 | 30
Years | 66.23 (13.31) | 58.17 (11.52)

3. Primary Outcome: Percentage of Patients With Accompanying Diseases
Description: At the beginning of the study, the patients were asked whether there were any of the following accompanying diseases and the percentage of patients with accompanying disease in both groups were recorded:
  * Diabetes mellitus
  * Hypertension
  * Coronary artery disease
  * Cardiac failure
  * Chronic obstructive pulmonary disease
  * Malignancy
  * Immunodeficiency
Time Frame: At the first day of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 30 | 30
Participants
  Diabetes Mellitus | 10 | 9
  Hypertension | 12 | 15
  Coronary artery disease | 8 | 5
  Cardiac failure | 1 | 0
  Chronic obstructive pulmonary disease | 3 | 6
  Malignancy | 1 | 0
  Immunodeficiency | 1 | 0

4. Primary Outcome: Percentage of Patients With Baseline Clinical Symptoms
Description: At the beginning of the study, the patients were asked whether there were any of the following clinical symptoms and the percentage of patients with any of the clinical symptoms in both groups were recorded:
  * Fever
  * Cough
  * Sore throat
  * Dispnea
  * Headache
  * Weakness
  * Myalgia
  * Diarrhea
  * Nausea or vomiting
Time Frame: At the first day of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 30 | 30
Participants
  Fever | 13 | 15
  Cough | 14 | 16
  Sore throat | 1 | 3
  dyspnea | 19 | 23
  Headache | 2 | 5
  Weakness | 11 | 13
  Myalgia | 7 | 9
  Diarrhea | 0 | 1
  Nausea or vomiting | 0 | 1

5. Primary Outcome: Body Temperature Means of the Patients
Description: At the beginning of the study, the body temperatures (as degree celcius) of the patients were measured and the mean body temperature values of both groups were recorded.
Time Frame: At the first day of the study
Measure: Mean (Standard Deviation); unit: Degree celcius
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 30 | 30
Degree celcius | 36.8 (0.8) | 36.9 (0.7)

6. Primary Outcome: Heart Rate Means of the Patients
Description: At the beginning of the study, the heart rates (as per minute) of the patients were measured and the mean heart rate values of both groups were recorded.
Time Frame: At the first day of the study
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 30 | 30
beats per minute | 92 (18) | 88 (12)

7. Primary Outcome: Respiratory Rate Means of the Patients
Description: At the beginning of the study, the respiratory rates (as per minute) of the patients were measured and the mean respiratory rate values of both groups were recorded.
Time Frame: At the first day of the study
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 30 | 30
breaths per minute | 24.7 (0.7) | 24 (5)

8. Primary Outcome: Systolic and Diastolic Pressure Means of the Patients
Description: At the beginning of the study, the systolic and diastolic pressures (as mmHg) of the patients were measured and the mean systolic and diastolic pressure values of both groups were recorded.
Time Frame: At the first day of the study
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 30 | 30
mmHg
  Systolic pressure | 124.61 (15.37) | 124.39 (15.60)
  Diastolic pressure | 73.43 (8.47) | 75.64 (9.79)

9. Primary Outcome: Number of Participants With Clinical Response
Description: The presence of at least two of the following criteria in patients at the end of 5th day were accepted as "clinical response": Extubation in mechanically ventilated patients, respiratory rate <26/min, SpO2 level in room air >90%, PaO2/FiO2 >300 in patients receiving oxygen, presence of at least two of the 2-point reduction criteria in "Sequential Organ Failure Assessment (SOFA)" score.
Time Frame: From starting to the end of ivermectin therapy (0 to the end of 5th day)
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 30 | 30
Participants | 11 | 14
Statistical Analysis 1: Comparison: Control Group vs Study Group; Test type: Superiority; p = 0.43, Chi-squared — A p<0.05 value was considered statistically significant

10. Primary Outcome: Changes in Oxygen Saturation (SpO2) Values
Description: Baseline SpO2 values of the patients were recorded in both groups. Then, their treatments were started and SpO2 values at the end of the 1st (TD1), 3rd (TD3) and 5th days (TD5) were also recorded. The end of the 5th day was accepted as the primary endpoint. While the change in SpO2 values on the 1st, 3rd and 5th days after the basal value calculated graphically, the change in the SpO2 value at the end of the 5th day (primary endpoint) with the baseline value was compared statistically (the results were given as p value).
Time Frame: From starting to the end of ivermectin therapy (0 to the end of 5th day)
Measure: Mean (Standard Deviation); unit: percentage of peripheral capillary O2
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 30 | 30
percentage of peripheral capillary O2
  Baseline | 89.67 (5.09) | 89.93 (6.51)
  TD1 | 90.50 (7.47) | 92.85 (4.86)
  TD3 | 91.90 (4.97) | 93.07 (4.12)
  TD5 | 93.00 (3.25) | 93.52 (4.36)
Statistical Analysis 1: Comparison: Control Group vs Study Group; Test type: Superiority; p = 0.14, Wilcoxon (Mann-Whitney) — A p<0.05 value was considered statistically significant

11. Primary Outcome: Changes in the Ratio of Partial Pressure of Oxygen (PaO2) to Fraction of Inspired Oxygen (FiO2) (PaO2/FiO2)
Description: Baseline PaO2/FiO2 ratios of the patients were recorded in both groups. Then, their treatments were started and PaO2/FiO2 ratios at the end of the 1st (TD1), 3rd (TD3) and 5th days (TD5) were also recorded. The end of the 5th day was accepted as the primary endpoint. While the change in PaO2/FiO2 ratios on the 1st, 3rd and 5th days after the basal ratio was calculated graphically, the change in the PaO2/FiO2 ratio at the end of the 5th day (primary endpoint) with the baseline value was compared statistically (the results were given as p value).
Time Frame: From starting to the end of ivermectin therapy (0 to the end of 5th day)
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 30 | 30
Ratio
  Baseline | 197.44 (102.31) | 158.83 (88.15)
  TD1 | 181.83 (99.62) | 147.31 (74.15)
  TD3 | 174.77 (94.74) | 147.74 (83.30)
  TD5 | 180.13 (95.43) | 178.94 (98.21)
Statistical Analysis 1: Comparison: Control Group vs Study Group; Test type: Superiority; p = 0.68, Wilcoxon (Mann-Whitney) — A p<0.05 value was considered statistically significant

12. Primary Outcome: Changes in Serum Lymphocyte Counts
Description: Baseline Serum Lymphocyte counts (cell/mm^3) of the patients were recorded in both groups. Then, their treatments were started and Serum Lymphocyte counts at the end of the 1st (TD1), 3rd (TD3) and 5th days (TD5) were also recorded. The end of the 5th day was accepted as the primary endpoint. While the change in Serum Lymphocyte counts on the 1st, 3rd and 5th days after the basal level was calculated graphically, the change in the Serum Lymphocyte count at the end of the 5th day (primary endpoint) with the baseline count was compared statistically (the results were given as p value).
Time Frame: From starting to the end of ivermectin therapy (0 to the end of 5th day)
Measure: Mean (Standard Deviation); unit: cell/mm^3
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 30 | 30
cell/mm^3
  Baseline | 1010 (438) | 932 (483)
  TD1 | 1034 (450) | 928 (607)
  TD3 | 977 (575) | 1021 (648)
  TD5 | 968 (477) | 1273 (822)
Statistical Analysis 1: Comparison: Control Group vs Study Group; Test type: Superiority; p = 0.15, Wilcoxon (Mann-Whitney) — A p<0.05 value was considered statistically significant

13. Primary Outcome: Changes in the Ratio of Polymorphonuclear Leukocyte Count to Lymphocyte Count (PNL/L)
Description: Baseline PNL/L ratio of the patients were recorded in both groups. Then, their treatments were started and PNL/L ratios at the end of the 1st (TD1), 3rd (TD3) and 5th days (TD5) were also recorded. The end of the 5th day was accepted as the primary endpoint. While the change in PNL/L ratios on the 1st, 3rd and 5th days after the basal level was calculated graphically, the change in the PNL/L ratio at the end of the 5th day (primary endpoint) with the baseline ratio was compared statistically (the results were given as p value).
Time Frame: From starting to the end of ivermectin therapy (0 to the end of 5th day)
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 30 | 30
Ratio
  Baseline | 7.48 (6.41) | 8.77 (8.35)
  TD1 | 7.74 (7.47) | 10.82 (8.55)
  TD3 | 9.26 (7.58) | 9.02 (13.08)
  TD5 | 9.88 (8.45) | 7.16 (4.97)
Statistical Analysis 1: Comparison: Control Group vs Study Group; Test type: Superiority; p = 0.37, Wilcoxon (Mann-Whitney) — A p<0.05 value was considered statistically significant

14. Primary Outcome: Changes in Serum Ferritin Levels
Description: Baseline serum ferritin levels (mg/dL) of the patients were recorded in both groups. Then, their treatments were started and serum ferritin levels at the end of the 1st (TD1), 3rd (TD3) and 5th days (TD5) were also recorded. The end of the 5th day was accepted as the primary endpoint. While the change in serum ferritin levels on the 1st, 3rd and 5th days after the basal level was calculated graphically, the change in the serum ferritin level at the end of the 5th day (primary endpoint) with the baseline level was compared statistically (the results were given as p value).
Time Frame: From starting to the end of ivermectin therapy (0 to the end of 5th day)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 30 | 30
mg/dL
  Baseline | 747.05 (800.54) | 682.75 (470.08)
  TD1 | 783.03 (827.10) | 834.94 (624.12)
  TD3 | 881.17 (779.95) | 875.90 (694.52)
  TD5 | 1028.24 (777.08) | 875.12 (1193.06)
Statistical Analysis 1: Comparison: Control Group vs Study Group; Test type: Superiority; p = 0.12, Wilcoxon (Mann-Whitney) — A p<0.05 value was considered statistically significant

15. Primary Outcome: Changes in Serum D-dimer Levels
Description: Baseline serum D-dimer levels (mg/L) of the patients were recorded in both groups. Then, their treatments were started and serum D-dimer levels at the end of the 1st (TD1), 3rd (TD3) and 5th days (TD5) were also recorded. The end of the 5th day was accepted as the primary endpoint. While the change in serum D-dimer levels on the 1st, 3rd and 5th days after the basal level was calculated graphically, the change in the serum D-dimer level at the end of the 5th day (primary endpoint) with the baseline level was compared statistically (the results were given as p value).
Time Frame: From starting to the end of ivermectin therapy (0 to the end of 5th day)
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 30 | 30
mg/L
  Baseline | 1.32 (2.04) | 1.25 (1.71)
  TD1 | 2.80 (5.66) | 1.40 (1.73)
  TD3 | 4.14 (9.91) | 3.24 (11.60)
  TD5 | 3.58 (8.27) | 5.85 (5.28)
Statistical Analysis 1: Comparison: Control Group vs Study Group; Test type: Superiority; p = 0.22, Wilcoxon (Mann-Whitney) — A p<0.05 value was considered statistically significant

16. Primary Outcome: Genetic Examination of Haplotypes and Mutations That Cause Function Losing for Ivermectin Metabolism
Description: A blood sample was taken from the patients included in the study group, after taking or during the first dose of ivermectin. From the blood samples, haplotypes and mutations that cause the function losing were investigated by performing sequence analysis of multidrug resistance 1 (MDR1)/ABCB1 and CYP3A4 genes with Sanger method. In case of detection of mutation, the patient were excluded from the study and if observed, side effects of ivermectin were noted.
Time Frame: At the first day of ivermectin therapy (1st day)
Population: We aimed to investigate the effectiveness/safety of adding ivermectin to the COVID-19 treatment in patients without mutation. Since ivermectin was not given to the control group, no blood sample was taken from these patients for mutation screening. The reason why there are 36 patients in the study group in this table is to indicate that there are 6 patients who were included in the study group but were removed from the study group because of a mutation and were replaced by additional patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 0 | 36
Participants
  Mutation positive | 0 | 6
  Mutation negative | 0 | 30

17. Primary Outcome: Treatment-Related Adverse Events as Assessed by CTCAE v4.0
Description: Adverse effects of ivermectin and drugs other than ivermectin (Hydroxychloroquine, favipiravir, azithromycin) were evaluated in the patients in the study group and and the number of participants were noted.
  Adverse effects of drugs other than ivermectin (Hydroxychloroquine, favipiravir, azithromycin) were evaluated in the patients in the control group and and the number of participants were noted.
Time Frame: At the first 5 days of study
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 30 | 30
Participants
  Nausea and vomiting | 2 | 0
  Increase in liver function tests | 1 | 0

18. Secondary Outcome: Number of Participants With Clinical Response
Description: The presence of at least two of the following criteria in patients on the 10th day were accepted as "clinical response": Respiration rate between 22-24/min, SpO2 level in room air >95%, absence of oxygen requirement, observation of radiological improvement in control lung tomography and no need for intensive care.
Time Frame: 10 days (5 days ivermectin therapy plus 5 days follow-up)
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 30 | 30
Participants | 16 | 22
Statistical Analysis 1: Comparison: Control Group vs Study Group; Test type: Superiority; p = 0.10, Chi-squared — A p<0.05 value was considered statistically significant

19. Secondary Outcome: Mortality
Description: The number of died patients were evaluated in study and control groups
Time Frame: Through study completion, an average of 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 30 | 30
Participants | 9 | 6
Statistical Analysis 1: Comparison: Control Group vs Study Group; Test type: Superiority; p = 0.37, Chi-squared — A p<0.05 value was considered statistically significant

20. Secondary Outcome: Changes in Oxygen Saturation (SpO2) Values
Description: In both groups, after the treatment period was completed (first 5 days, primary endpoint), patients were followed up for 5 more days (follow-up period). SpO2 values at the end of 6th (FD1), 8th (FD3) and 10th day (FD5) were also recorded. The end of the 10th day was accepted as the secondary endpoint. While the change in SpO2 values on the 6th, 8th and 10th days was calculated graphically, the change in the SpO2 value at the end of the 10th day (secondary endpoint) with the baseline value was compared statistically (the results were given as p value).
Time Frame: From 6th to the end of 10th day
Measure: Mean (Standard Deviation); unit: percentage of peripheral capillary O2
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 30 | 30
percentage of peripheral capillary O2
  Baseline | 89.67 (5.09) | 89.93 (6.51)
  FD1 | 92.43 (2.86) | 94.54 (2.21)
  FD3 | 92.91 (2.71) | 94.24 (2.76)
  FD5 | 93.00 (3.93) | 95.35 (2.72)
Statistical Analysis 1: Comparison: Control Group vs Study Group; Test type: Superiority; p = 0.03, Wilcoxon (Mann-Whitney) — A p<0.05 value was considered statistically significant

21. Secondary Outcome: Changes in the Ratio of Partial Pressure of Oxygen (PaO2) to Fraction of Inspired Oxygen (FiO2) (PaO2/FiO2)
Description: In both groups, after the treatment period was completed (first 5 days, primary endpoint), patients were followed up for 5 more days (follow-up period). PaO2/FiO2 ratios at the end of 6th (FD1), 8th (FD3) and 10th day (FD5) were also recorded. The end of the 10th day was accepted as the secondary endpoint. While the change in PaO2/FiO2 ratios on the 6th, 8th and 10th days was calculated graphically, the change in the PaO2/FiO2 ratio at the end of the 10th day (secondary endpoint) with the baseline ratio was compared statistically (the results were given as p value).
Time Frame: From 6th to the end of 10th day
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 30 | 30
Ratio
  Baseline | 197.44 (102.31) | 158.83 (88.15)
  FD1 | 204.28 (109.51) | 199.83 (85.02)
  FD3 | 211.75 (127.62) | 227.43 (103.71)
  FD5 | 220.78 (127.26) | 236.33 (85.66)
Statistical Analysis 1: Comparison: Control Group vs Study Group; Test type: Superiority; p = 0.39, Wilcoxon (Mann-Whitney) — A p<0.05 value was considered statistically significant

22. Secondary Outcome: Changes in Serum Lymphocyte Counts
Description: In both groups, after the treatment period was completed (first 5 days, primary endpoint), patients were followed up for 5 more days (follow-up period). Serum lymphocyte counts (cell/mm^3) at the end of 6th (FD1), 8th (FD3) and 10th day (FD5) were also recorded. The end of the 10th day was accepted as the secondary endpoint. While the change in serum lymphocyte counts on the 6th, 8th and 10th days was calculated graphically, the change in the serum lymphocyte count at the end of the 10th day (secondary endpoint) with the baseline value was compared statistically (the results were given as p value).
Time Frame: From 6th to the end of 10th day
Measure: Mean (Standard Deviation); unit: cell/mm^3
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 30 | 30
cell/mm^3
  Baseline | 1010 (438) | 932 (483)
  FD1 | 916 (411) | 1403 (869)
  FD3 | 1086 (880) | 1668 (819)
  FD5 | 1256 (710) | 1698 (1438)
Statistical Analysis 1: Comparison: Control Group vs Study Group; Test type: Superiority; p = 0.24, Wilcoxon (Mann-Whitney) — A p<0.05 value was considered statistically significant

23. Secondary Outcome: Changes in the Ratio of Polymorphonuclear Leukocyte Count to Lymphocyte Count (PNL/L)
Description: In both groups, after the treatment period was completed (first 5 days, primary endpoint), patients were followed up for 5 more days (follow-up period). PNL/L ratios at the end of 6th (FD1), 8th (FD3) and 10th day (FD5) were also recorded. The end of the 10th day was accepted as the secondary endpoint. While the change in PNL/L ratios on the 6th, 8th and 10th days was calculated graphically, the change in the PNL/L ratio at the end of the 10th day (secondary endpoint) with the baseline value was compared statistically (the results were given as p value).
Time Frame: From 6th to the end of 10th day
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 30 | 30
Ratio
  Baseline | 7.48 (6.41) | 8.77 (8.35)
  FD1 | 10.49 (7.10) | 6.90 (11.84)
  FD3 | 9.66 (10.99) | 5.81 (9.99)
  FD5 | 6.19 (4.85) | 7.34 (8.09)
Statistical Analysis 1: Comparison: Control Group vs Study Group; Test type: Superiority; p = 0.56, Wilcoxon (Mann-Whitney) — A p<0.05 value was considered statistically significant

24. Secondary Outcome: Changes in Serum Ferritin Levels
Description: In both groups, after the treatment period was completed (first 5 days, primary endpoint), patients were followed up for 5 more days (follow-up period). Serum ferritin levels (mg/dL) at the end of 6th (FD1), 8th (FD3) and 10th day (FD5) were also recorded. The end of the 10th day was accepted as the secondary endpoint. While the change in serum ferritin levels on the 6th, 8th and 10th days was calculated graphically, the change in the serum ferritin level at the end of the 10th day (secondary endpoint) with the baseline value was compared statistically (the results were given as p value).
Time Frame: From 6th to the end of 10th day
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 30 | 30
mg/dL
  Baseline | 747.05 (800.54) | 682.75 (470.08)
  FD1 | 1076.88 (704.05) | 628.45 (580.10)
  FD3 | 1097.57 (595.22) | 433.48 (641.82)
  FD5 | 1206.90 (782.84) | 494.71 (349.78)
Statistical Analysis 1: Comparison: Control Group vs Study Group; Test type: Superiority; p = 0.005, Wilcoxon (Mann-Whitney) — A p<0.05 value was considered statistically significant

25. Secondary Outcome: Changes in Serum D-dimer Levels
Description: In both groups, after the treatment period was completed (first 5 days, primary endpoint), patients were followed up for 5 more days (follow-up period). Serum D-dimer levels (mg/L) at the end of 6th (FD1), 8th (FD3) and 10th day (FD5) were also recorded. The end of the 10th day was accepted as the secondary endpoint. While the change in Serum D-dimer levels on the 6th, 8th and 10th days was calculated graphically, the change in the serum D-dimer level at the end of the 10th day (secondary endpoint) with the baseline value was compared statistically (the results were given as p value).
Time Frame: From 6th to the end of 10th day
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 30 | 30
mg/L
  Baseline | 1.32 (2.04) | 1.25 (1.71)
  FD1 | 3.45 (6.60) | 1.37 (2.53)
  FD3 | 1.63 (1.38) | 0.89 (2.45)
  FD5 | 1.49 (2.28) | 0.71 (0.96)
Statistical Analysis 1: Comparison: Control Group vs Study Group; Test type: Superiority; p = 0.03, Wilcoxon (Mann-Whitney) — A p<0.05 value was considered statistically significant

26. Secondary Outcome: Rate of COVID-19 Polymerase Chain Reaction (PCR) Test Negativity
Description: At the end of the follow-up period (10th day), patients in the study and control group were investigated by PCR test for SARS-CoV-2 and the negative results were recorded as percentage for both groups.
Time Frame: At the end of 10th day
Population: PCR test was applied to 8 patients in the control group and 16 patients in the study group at the end of the study (secondary endpoint).
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 8 | 16
Participants | 3 | 14
Statistical Analysis 1: Comparison: Control Group vs Study Group; Test type: Superiority; p = 0.01, Chi-squared — A p<0.05 value was considered statistically significant

27. Secondary Outcome: Treatment-Related Adverse Events as Assessed by CTCAE v4.0
Description: as for outcome 17
Time Frame: From the 6th day of study to the 10th day of study
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 30 | 30
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From the beginning of the study to the end of the 10th day
Description: In our study, it was also aimed to detect mutations that impair ivermectin metabolism and report side effects that may occur due to these mutations, and these mutations were detected in 6 patients initially included in the study group. Since these patients were excluded from the study on the first day following the mutation detection and their ivermectin treatment was discontinued, they were evaluated separately from the other patients included in the study.
Groups:
- Participants With Mutations: Patients that were included in the study group and excluded from the study because one or both of the multidrug resistance 1 (MDR1) / ABCB1 and CYP3A4 genes were detected in the blood sample taken at the beginning of ivermectin treatment on the first day
Arm/Group | Control Group | Study Group | Participants With Mutations
All-Cause Mortality (participants affected / at risk) | 9/30 | 6/30 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 5/6
Other Adverse Events (participants affected / at risk) | 3/30 | 0/30 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control Group (N=30) | Study Group (N=30) | Participants With Mutations (N=6)
Encephalopathy (Nervous system disorders) | 0 | 0 | 5
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=30) | Study Group (N=30) | Participants With Mutations (N=6)
Nausea and vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Increase in liver function tests (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-04-05): https://cdn.clinicaltrials.gov/large-docs/09/NCT04646109/Prot_000.pdf
  • Informed Consent Form (2020-04-05): https://cdn.clinicaltrials.gov/large-docs/09/NCT04646109/ICF_001.pdf
  • Statistical Analysis Plan (2020-04-05): https://cdn.clinicaltrials.gov/large-docs/09/NCT04646109/SAP_002.pdf